CLINICAL TRIAL: NCT03277300
Title: Enteral and Parenteral Feeding in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelhamid, doctor, Assiut University
Other Study IDs: EN&PN
Record Dates: First submitted 2017-08-28; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: dietary supplement — good dietary supplement for critically ill patients

SUMMARY:
Supplementation of insufficient enteral nutrition with parenteral nutrition may optimize nutritional support and avert negative energy balance in critically ill patients, thereby improving outcome.

DETAILED DESCRIPTION:
Malnutrition is a common and serious problem in intensive care units. Negative energy balance has been associated with increased morbidity and mortality in critically ill patients. The increased incidence of complications related to malnutrition correlates with increased length of hospital stay and overall health care costs. Although early enteral nutrition is the preferred method of feeding critically ill patients, enteral nutrition alone often fails to supply adequate calories and nutrients to critically ill patients, who are frequently hypermetabolic.

Artificial nutrition support has evolved into a primary therapeutic intervention to prevent metabolic deterioration and loss of lean body mass with the aim to improve the outcome of critically ill patients. Apart from the timing of initiation and the targeted amount of macronutrients, the route of delivery is viewed as an important determinant of the effect of the nutritional intervention.

Using the enteral route is considered to be more physiologic, providing nutritional and various non-nutritional benefits including maintenance of structural and functional gut integrity as well as preserving intestinal microbial diversity.

The disadvantage of enteral nutrition is related to a potential lower nutritional adequacy particularly in the acute disease phase and in the presence of gastrointestinal dysfunction.

In contrast, parenteral nutrition may better secure the intended nutritional intake but is associated with more infectious complications, most likely due to hyperalimentation and hyperglycemia.

Supplementation of insufficient enteral nutrition with parenteral nutrition may optimize nutritional support and avert negative energy balance in critically ill patients, thereby improving outcome.

Combining parenteral nutrition with enteral nutrition constitutes a strategy to prevent nutritional deficit but may increase risk of overfeeding, which has been associated with liver dysfunction, infection, and prolonged ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to CCU (critical care unit)who are in need for either enteral or parenteral during duration of the study will be included

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data will be collected and analyzed using SPSS version 20. Normally distributed data will be expressed in form of mean and SD while not normally distributed data will be expressed in form of median and range. Nominal data will be expressed in form of frequency (percentage). P value will be significant if < 0.05.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
ts Overall mortality | one year
  Determined by hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: NoorEldeen AbdElazeem, professor, Study Chair — Assiut University

REFERENCES:
- [Background] DerSimonian R, Laird N. Meta-analysis in clinical trials. Control Clin Trials. 1986 Sep;7(3):177-88. doi: 10.1016/0197-2456(86)90046-2. PMID 3802833
- [Background] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094